CLINICAL TRIAL: NCT06386926
Title: Radial Shockwave Versus Ultrasound Phonophoresis in Management of Chronic Supraspinatus Tendinitis
Brief Title: Radial Shockwave Versus Ultrasound Phonophoresis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shady Bahaaldin Alkadry, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005075
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Supraspinatus Tendinitis
Keywords: Shockwave , phonophoresis , supraspinatus tendinitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): 23 subjects will Receive radial shockwave by ( Storz Medical /SN:BS.3517 ) for 3 sessions one session per week for four consecutive weeks and conventional physical therapy
  Interventions: Other: Electro Therapy
- Experimental group 2 (Experimental): 23 subjects will receive Ultrasound phonophoresis using diclofenac Na+( voltaren) by ( Sonopuls 490 / SN : 36 602 ) for 12 session, 3 sessions per week and same conventional physical therapy
  Interventions: Other: Electro Therapy
- Control group (Other): 23 subjects will receive conventional physical therapy modalities in the for 3 sessions per week for 4 weeks in form of Stretching Exercise in form of exercise of posterior shoulder capsule, strengthening exercises all have been recommended as essential for any shoulder rehabilitation program. These exercise include shoulder flexion, scaption.
  ,Tens applied for 20 minutes per session using (Enraf Nonius (Endomed 482) SN : 36853 )
  Interventions: Other: Electro Therapy

INTERVENTIONS:
Other: Electro Therapy — radial shockwave 3 sessions one session per week for four consecutive weeks ,receive Ultrasound phonophoresis using diclofenac Na+ 12 session, 3 sessions per week and conventional physical therapy modalities in the form of 3 sessions every week for 8 weeks

SUMMARY:
Comparative study to compare the effect of radial shockwave versus ultrasound phonophoresis in management of chronic supraspinatus tendinitis consists of 3 groups exp1(shockwave treatment + conventional physical therapy) , exp2( ultrasound phonophoresis+ conventional physical therapy) and control group ( conventional physical therapy)

ELIGIBILITY:
Inclusion Criteria:- BMI 18.5-24.9

* 18 years to 60
* with Unilateral Chronic Supraspinatus Tendinitis.
* Tenderness is found over the supraspinatus as it passes sub-acrominal and anterolateral.
* The patient reported with positive Jobe's test (empty can test)
* The patient reported pain with active shoulder elevation in the scapular plane (eg: welders, plate workers, slaughterhouse workers and overhead playing athletes).
* The patient reported pain with resisted isometric abduction

Exclusion Criteria:

* Case reports, treatments after surgery, did not meet our specified outcome parameters, traumatic incidents,
* Partial tears at surgery
* Massive retracted tears at surgery
* Frozen shoulder.
* Rotator cuff tear.
* Glenohumeral or acromioclavicular arthritis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
change in the thickness of supraspinatus tendon | before start of treatment and 4 weeks following end of treatment
  Ultrasonography
change in pain intesity | before start of treatment and 4 weeks following end of treatment , score from 0-10 ,0=no pain , 10= unbearable pain
  VAS ( visual analog scale score)
Change in shoulder range of motion | before start of treatment and 4 weeks following end of treatment
  electro goniometer

SECONDARY OUTCOMES:
Function of the Upper Limb | before start of treatment and 4 weeks following end of treatment, it measure the disability/symptom section (11 items, scored 1-5)
  Quick DASH Questionnaire score
measure weight in kg and height in cm | before starting the assessment
  Weight and height scale for determining BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided